CLINICAL TRIAL: NCT00374543
Title: Ziprasidone for the Treatment of Generalized Anxiety Comorbidity in Patients With Bipolar Disorder
Brief Title: Ziprasidone for the Treatment of Generalized Anxiety in Patients With Bipolar Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment goal could not be achieved
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Naomi M. Simon, Director, Center for Anxiety and Traumatic Stress Disorders, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-P-000142
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Generalized Anxiety Disorder; Bipolar Disorder
Keywords: Bipolar Disorder; Generalized Anxiety Disorder; Double-blind; Placebo-controlled; Ziprasidone
MeSH Terms: conditions — Generalized Anxiety Disorder; Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ziprasidone (Experimental): Ziprasidone will be dosed on a twice daily (BID) basis, with flexible dosing based on tolerability, with a total daily dose in the range of 40 to 160 mg/day, for 8 weeks. This time period reflects the rapid onset of effect seen in studies of atypical antipsychotics, but allows time for a potentially longer response for some anxiety symptoms.
  Interventions: Drug: Ziprasidone
- Placebo Capsules (Placebo Comparator): Identical placebo capsules will be dosed on a BID basis, with flexible dosing based on tolerability, with a total daily dose in the range of 40 to 160 mg/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziprasidone — Ziprasidone, flexibly dosed from 40 to 160 mg/day, for 8 weeks.
  Other Names: Geodon
  Arms: Ziprasidone
Drug: Placebo — Placebo administered daily for 8 weeks
  Other Names: Control
  Arms: Placebo Capsules

SUMMARY:
This study proposes to examine the potential safety and efficacy of ziprasidone for patients with anxiety and bipolar disorder on anxiety outcomes, bipolar symptoms, and on measures of quality of life and resilience.

DETAILED DESCRIPTION:
This study would be the first prospective, placebo-controlled study to our knowledge of any pharmacotherapy strategy for the treatment of comorbid generalized anxiety (or any comorbid anxiety) in patients with bipolar disorder. Our hypotheses are:

1. Ziprasidone flexibly dosed from 40 to 160 mg/day will reduce anxiety symptoms significantly more than placebo in patients with bipolar disorder who have a full or subsyndromal diagnosis of generalized anxiety disorder (GAD).
2. Ziprasidone will be well tolerated in patients with generalized anxiety based on the incidence of treatment emergent adverse effects during 8 weeks of therapy, and based on a lack of worsening of bipolar depression, mania or hypomania compared to placebo.
3. Treatment with ziprasidone will have a significantly greater positive impact on measures of quality of life and resilience than placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, aged 18 to 75 years.
* Diagnosis of Bipolar Disorder (Bipolar I or Bipolar II).
* Current diagnosis of Generalized Anxiety Disorder (GAD).
* Participants must be on at least one of the following mood stabilizers at steady dose for at least 4 weeks prior to randomization: lithium with blood levels between 0.4-1.4 meq/L, valproic acid/divalproate sodium (with levels between 50-150 ugm/dl) carbamazepine (blood levels between 4-12 mcg/ml), or lamotrigine (dosed 50-400 mg/day).

Exclusion Criteria:

* Pregnant or lactating women or others not using acceptable means of birth control (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, implanted progesterone rods stabilized for at least 3 months).
* Patients with current or history of schizophrenia, or patients with current mania, hypomania at study entry. Lifetime psychosis and dementia are exclusionary.
* Patients with current obsessive-compulsive disorder or posttraumatic stress disorder are excluded.
* Patients with a history of alcohol or substance abuse or dependence within the last three months.
* Patients with significant unstable medical illness likely to result in hospitalization or acute medical care. In addition, patients with an established diagnosis of diabetes mellitus are excluded.
* Current cognitive behavioral therapy directed toward the treatment of generalized anxiety disorder.
* History of hypersensitivity to or lack of response to ziprasidone.
* Concomitant treatment with other typical or atypical antipsychotics; patients should be off other typical or atypical antipsychotics for at least one week prior to study baseline.
* Patients with significant suicidal ideation or who have enacted suicidal behaviors within 3 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
* Patients who have had a psychiatric hospitalization (including for bipolar disorder) in the past 3 months are excluded.
* Seizure disorders with the exception of a history of febrile seizures if they occurred during childhood, were isolated, and did not recur in adulthood.
* History of Neuroleptic Malignant Syndrome.
* Individuals with current clinically significant orthostatic hypotension are excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M. Simon, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Anxiety and Traumatic Stress Disorders at Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Numerous attempts were made to increase enrollment since study inception. Researchers made use of Radio, Internet and print ads, as well as weekly Internet postings. Researchers also circulated an IRB-approved GAD checklist in a Bipolar Clinic waiting area in order to increase enrollment and recruit a clinically relevant sample.
Pre-assignment Details: A total of thirteen individuals signed consent, but only three were randomized to the study arms. The other ten participants were excluded from the study for meeting various exclusion criteria.
Groups:
- Ziprasidone, 40 to 160 mg/Day: Patients with Bipolar Disorder and Anxiety Comorbidity who consent and meet entry criteria will be randomized to placebo or Ziprasidone. Ziprasidone will be dosed on a BID basis, with flexible dosing based on tolerability, with a total daily dose in the range of 40 to 160 mg/day.
- Placebo: Patients with Bipolar Disorder and Anxiety Comorbidity who consent and meet entry criteria will be randomized to placebo or Ziprasidone. Identical placebo capsules will be dosed on a BID basis, with flexible dosing based on tolerability, with a total daily dose in the range of 40 to 160 mg/day.
Period: Overall Study
Arm/Group | Ziprasidone, 40 to 160 mg/Day | Placebo
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone, 40 to 160 mg/Day | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0
  >= 18 to 75 years | 2 | 1 | 3
  >75 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I)
Description: A secondary categorical outcome of response will be defined as a Clinical Global Impression Improvement Score (CGI-I) of 1 or 2. The CGI-I is a 7 point clinician-rated scale that assesses symptom improvement or worsening relative to a previous assessment. Lower ratings reflect greater improvement.
  Due to study termination, there are not results for primary and secondary outcome measures.
Time Frame: 8 weeks
Reporting Status: Not Posted

2. Primary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: The 14-item Hamilton Anxiety Rating Scale (HAM-A) (Hamilton, 1959) was developed to assess anxiety in a clinical population. It is considered a measure of general anxiety across anxiety disorders, in addition to being a gold standard measure for GAD.
  Due to study termination, there are not results for primary and secondary outcome measures.
Time Frame: 8 weeks
Population: Zero participants were analyzed because recruitment was very low. Due to this, we felt any analysis done would not be usable for accurate analyses.
Arm/Group | Ziprasidone, 40 to 160 mg/Day | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ziprasidone, 40 to 160 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziprasidone, 40 to 160 mg/Day (N=2) | Placebo (N=1)
Tremulousness (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Urinary Hesitancy (General disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 1 (3) | 0 (0)
Akathisia (General disorders) | 1 (2) | 0 (0)
Jitteriness (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated due to extreme difficulties in participant recruitment. Therefore, the sample size is extremely low, leaving inconclusive data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No